CLINICAL TRIAL: NCT03424174
Title: Clinical Outcome and Cytokine Expression in Blood After Coated in Comparison to Uncoated TKA
Brief Title: Clinical Outcome and Cytokine Expression After TKA
Acronym: TKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKA cytokine
Record Dates: First submitted 2016-03-17; First posted 2018-02-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis
Keywords: TKA, cytokine, coating
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Coated Total Knee Arthroplasty (Experimental): Implantation coated Total Knee Arthroplasty
  Interventions: Device: Coated Total Knee Arthroplasty
- Standard Total Knee Arthroplasty (Active Comparator): Implantation Standard Total Knee Arthroplasty
  Interventions: Device: Standard Total Knee Arthroplasty

INTERVENTIONS:
Device: Coated Total Knee Arthroplasty — Implantation coated Total Knee Arthroplasty
  Arms: Coated Total Knee Arthroplasty
Device: Standard Total Knee Arthroplasty — Implantation StandardTotal Knee Arthroplasty
  Arms: Standard Total Knee Arthroplasty

SUMMARY:
Comparison of coated and uncoated TKA with regard to cytokine expression and clinical results

DETAILED DESCRIPTION:
Comparison of coated and uncoated TKA with regard to cytokine expression and clinical results at 3 months, 1 year and 3 years after surgery

ELIGIBILITY:
Inclusion Criteria:

* Primary and secondary osteoarthritis
* understanding of german language

Exclusion Criteria:

* necessity of constrained TKA
* existence of other joint implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
cytokine expression | pre-op, 1 and 3 years post-op
  Changes of cytokine expression 1 and 3 years after surgery compared to pre-op

SECONDARY OUTCOMES:
Function assessed with Knee Society Score | pre-op, 3 months, 1 and 3 years post-op
  Knee Society Score (0 - 100 points, best 100)
Patient reported outcome assessed with Oxford Knee Score | pre-op, 3 months, 1 and 3 years post-op
  Oxford Knee Score (0 - 48 points, best 48)
Quality of life assessed with EQ 5D | pre-op, 3 months, 1 and 3 years post-op
  EQ 5D Index (0 - 1.0, best 1.0)
Activity assessed with UCLA activity score | pre-op, 3 months, 1 and 3 years post-op
  UCLA activity score (0 - 10 points, best 10)

OTHER OUTCOMES:
adverse events | 3 month, 1 year and 3 years post-op
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Lützner, MD, Principal Investigator — University Center of Orthopaedics and Traumatology, University Medicine Carl Gustav Carus Dresden
Locations (1):
- University Center of Orthopaedics and Traumatology, University Medicine Carl Gustav Carus Dresden, TU Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tille E, Beyer F, Lutzner C, Postler A, Thomas P, Summer B, Lutzner J. No difference in patient reported outcome and inflammatory response after coated and uncoated total knee arthroplasty - a randomized controlled study. BMC Musculoskelet Disord. 2023 Dec 14;24(1):968. doi: 10.1186/s12891-023-07061-x. PMID 38098024